CLINICAL TRIAL: NCT03611738
Title: Phase I Study of Ceritinib Plus Docetaxel in ALK-Negative, EGFR WT Advanced NSCLC
Brief Title: Ceritinib Plus Docetaxel in ALK-Negative, EGFR WT Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19656
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer; Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Stage IIIB; Stage IV Non-small Cell Lung Cancer; EGFR Negative Non-Small Cell Lung Cancer
Keywords: Advanced NSCLC; Advanced Non-small Cell Lung Cancer; anaplastic lymphoma kinase (ALK); ALK-negative; epidermal growth factor receptor (EGFR); wild-type (WT)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ceritinib; Tyrosine Kinase Inhibitors; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I Dose Escalation (Experimental): The design will recruit participants in cohorts of three patients each and will not allow for dose-skipping during escalation. A maximum of 18 participants will be enrolled for the phase I dose escalation. Three ceritinib dose levels have been identified for dose escalation (150 mg, 300 mg, and 450 mg), plus docetaxel at 75 mg. A backup dose (ceritinib 150 mg with docetaxel at 60 mg) is also prepared in case the three dose levels are too toxic. Therefore, four potential dose levels will be used for determination of maximum tolerated dose (MTD). The first cohort will start at dose level 1 (ceritinib 150 mg with docetaxel at 75 mg).
  Level -1 Backup Cohort: 150 mg ceritinib; 60 mg/m^2 docetaxel Level 1 Starting Cohort: 150 mg ceritinib; 75 mg/m^2 docetaxel Level 2 Cohort: 300 mg ceritinib; 75 mg/m^2 docetaxel Level 3 Cohort: 450 mg ceritinib; 75 mg/m^2 docetaxel
  Interventions: Drug: Ceritinib; Drug: Docetaxel
- Phase Ib Dose Expansion (Experimental): Treatment at recommended dose. Investigators plan to have 30 patients for the expansion cohort. This will include participants from the dose escalation portion receiving the recommended dose.
  Interventions: Drug: Ceritinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Ceritinib — Ceritinib daily by mouth (PO) with food, according to the dosage schedule outlined in the treatment arm.
  Other Names: Zykadia®; tyrosine kinase inhibitor
Drug: Docetaxel — Docetaxel intravenously (IV) every 3 weeks, according to the dosage schedule outlined in the treatment arm.
  Other Names: Taxotere®; intravenous microtubule inhibitor

SUMMARY:
The main purpose of this study is to find out what effects (good and bad) ceritinib (Zykadia®) used in combination with docetaxel (Taxotere®) will have on participants and their cancer. The results will help to determine the best safe dose of the combination of the medications Ceritinib (Zykadia®) and docetaxel (Taxotere®) and to find out if this combination of drugs will help people that have this type of Non-small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
In this phase I/IB clinical trial, participants with non-small cell lung cancer (NSCLC) who have progressed on prior platinum-based chemotherapy (maximum number of prior distinct regimens = 2) and are anaplastic lymphoma kinase (ALK)-negative/epidermal growth factor receptor (EGFR) wild-type (WT) will receive a combination of ceritinib and docetaxel.

Study rationale is that targeting ALK- and EGFR-negative lung tumors with ceritinib and microtubule inhibitors results in synergistic antitumor effects. Therefore, treatment with ceritinib and docetaxel is a rational combination.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide informed consent.
* Willingness and ability to comply with scheduled study visits and procedures.
* Adult men or women age ≥ 18 years.
* Histologic or cytologic diagnosis of advanced/metastatic Non-small Cell Lung Cancer (NSCLC), stage IIIB/IV.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 1 - 3 (no more than three) prior regimens for stage IIIB/IV disease, with at least one prior regimen (for any stage) containing a platinum-based agent. One prior PD-1 or PD-L1 antibody-based regimen is allowable and counts as a prior regimen. Prior therapy with a taxane is allowed.
* Participants enrolled on the phase 1b expansion portion of the trial must be willing and able to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 3 months prior to initiation of treatment on Day 1, and must be obtained after most recent tumor progression. Participants for whom newly-obtained samples cannot be provided (e.g., inaccessible or participant safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Prior radiation is allowed if patients have recovered from side effects.
* Potential participants with a prior history of brain metastases are eligible, provided:

  * The brain metastases have been treated
  * The patient is asymptomatic from the brain metastases
  * Corticosteroids prescribed for the management of brain metastases have been discontinued at least 7 days before registration to study
  * The brain metastases are stable on pre-registration imaging
  * There is no evidence of leptomeningeal disease
* Measurable metastatic disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Life expectancy > 3 months.
* Must have adequate organ and marrow function.
* Must have adequate laboratory values.
* Participants of child bearing potential must not be pregnant and must use established contraceptive strategies as outlined in the study protocol.

Exclusion Criteria:

* Rearrangements in ALK.
* Activating mutations in EGFR.
* Potential participants with active malignancies other than NSCLC, or prior curatively treated malignancy at high risk of relapse during the study period with the exception of localized squamous or basal cell skin cancers.
* Pregnant or breast feeding.
* Known hypersensitivity to ceritinib, docetaxel, or any of their excipients.
* Serious uncontrolled medical disorder, psychiatric condition or laboratory abnormalities that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Has had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior to starting study treatment or has not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy are exceptions and patients can receive study treatment ≥1 week after these procedures.
* A history of clinically significant noninfectious interstitial pneumonitis (i.e., limiting activities of daily living or requiring therapeutic intervention), including clinically significant radiation pneumonitis.
* Residual toxicity from prior anticancer therapy of grade 3 or greater (CTCAE v5.0), with the exception of alopecia
* Concurrent use of other anticancer approved or investigational agents within 2 weeks of the first dose of study treatment.
* In taxane pretreated patents, any history of dose-limiting toxicity with prior taxane therapy.
* A clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months).
* Uncontrolled diabetes mellitus, defined as fasting plasma glucose > 200 mg/dL.
* Impaired gastrointestinal (GI) function or GI disease that may alter absorption of ceritinib, or inability to swallow capsules
* Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with ceritinib and for the duration of participation:

  * Medication with a known risk of prolonging QT interval or inducing Torsades de Pointes
  * Strong inhibitors or strong inducers of CYP3A4/5 (see Appendix A for list)
  * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, and/or CYP2C9
  * Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (e.g., dabigatran, rivaroxaban, apixaban)
  * Enzyme-inducing anticonvulsive agents
  * Herbal medications, including but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | Up to 6 months
  Maximum tolerated dose corresponding to a risk of dose limiting toxicity (DLT) occurring in 30% of patients.
Phase Ib: Overall Response (OR) | Up to 30 months
  OR: Defined as the participant being alive and the tumor size evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 on subsequent imaging assessment consistent with a complete response (CR) or partial response (PR). Overall response rates will be calculated with a 2-sided 95% confidence interval (CI). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm (< 1 cm). Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 30 months
  PFS: Defined as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, will be summarized with the Kaplan-Meier curve. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm). (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Overall Survival (OS) | Up to 30 months
  OS: Defined as the time from study entry to death due to any cause, will be summarized with the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Saltos, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Advent Health Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida